CLINICAL TRIAL: NCT02209935
Title: RCT Early Rehabilitation Protocol vs. Usual Care in the Pediatric ICU for Children With Acute Brain Injury
Brief Title: RCT: Early Rehabilitation Protocol vs. Usual Care in the Pediatric ICU for Children With Acute Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Ericka Fink, Associate Professor, Pediatric Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCORI APDTO
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Pediatric Acute Neurologic Disease, Traumatic and Non-traumatic
Keywords: pediatric; acute neurologic disease; critical care; rehabilitation; outcome

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Typically, usual care is when therapies are not initiated until the treating team places an order for each element of care (physical, occupational, speech, and emotional therapy consultation).
  Interventions: Other: Usual care
- Early Rehabilitation Protocol (Experimental): Physical, occupational, speech, and emotional evaluation and support personalized to the subject's severity of illness and developmental status.
  Interventions: Other: Early Rehabilitation Protocol

INTERVENTIONS:
Other: Early Rehabilitation Protocol
  Arms: Early Rehabilitation Protocol
Other: Usual care
  Arms: Usual Care

SUMMARY:
Background. Early rehabilitation programs (ERP) that include physical, occupational, and speech therapies lessens debilitation and promotes return to previous physical and cognitive functioning and have been successfully applied in adult intensive care units (ICUs). Despite the fact that critically ill children with acute brain injury (ABI) are at increased risk of life-long disability and stunted development, benefits of ERP for this group have not been studied and are not standard of care in pediatric ICUs.

Objectives. The aims of this study are 1) To better understand current practices and barriers to use of these therapies and 2) To subsequently evaluate ERP vs. usual care in children with ABI in the ICU by randomizing children to these groups and measuring outcomes. We expect that ERP therapies are underutilized in the PICU and that outcomes in the ERP group will be superior compared to the usual care group.

Methods. The first task of this research program is to survey healthcare professionals (physicians, nurses, allied health) and families of children in the ICU about their hospital's resources, current practices, and barriers to ERP. This survey will be distributed to the 78 sites affiliated with the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI), a group of clinicians and researchers dedicated to improving child outcomes from critical illness. Next, we will enroll 175 children with ABI in a randomized, controlled trial of ERP versus usual care. Children enrolled in ERP will begin therapies by 48 hours of ICU admission and those in the usual care group will begin therapies when these services are ordered by treating physicians. Children aged 3-17 years with ABI expected to be admitted to the ICU > 48 hours due to trauma, infection, low oxygen, or low blood flow to the brain are eligible. Therapy interventions are individualized for the child's clinical status. The effectiveness of ERP will be measured using the Vineland Behavior Adaptive Scale (VABS) pre-ABI and 6 months post-ABI. This test, validated for children, assesses a child's physical and cognitive function as well as behavior. Other tests will be performed that assesses child and family quality of life and length of hospital admission. Our outcome tests were chosen because 1) They are the most important outcomes to families of children as surveyed in our ICU and 2) They are outcomes that can be influenced by ERP.

Summary. This is the first and largest study designed to evaluate whether ERP improves outcomes for critically ill children with ABI. We anticipate that rehabilitation practices in ICUs will be unprotocolized and under-utilized. We expect that patients in the ERP group will have superior adaptive and quality of life outcomes, outcomes important to families, without increasing adverse events compared to patients in the usual care group.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-17 years
* ABI due to TBI, ischemia, CNS infection / inflammation (i.e., meningitis, encephalitis), or cardiac arrest
* Subjects will be enrolled prior to 48 hours of PICU admission, have English or Spanish speaking parents/guardians, and en expected ICU stay ≥ 3 days

Exclusion Criteria:

* Children with a do not resuscitate status
* Pediatric Cerebral Performance Category (PCPC) score 4-5 (4=severe disability and 5=persistent vegetative state) prior to ABI or are not expected to survive > 24 hours will be excluded

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Vineland Adaptive Behavioral Scale score | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Piva TC, Ferrari RS, Schaan CW. Early mobilization protocols for critically ill pediatric patients: systematic review. Rev Bras Ter Intensiva. 2019 Jun 10;31(2):248-257. doi: 10.5935/0103-507X.20190038. PMID 31215603
- [Derived] Treble-Barna A, Beers SR, Houtrow AJ, Ortiz-Aguayo R, Valenta C, Stanger M, Chrisman M, Orringer M, Smith CM, Pollon D, Duffett M, Choong K, Watson RS, Kochanek PM, Fink EL; PICU-Rehabilitation Study Group, Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network, and Prevalence of Acute critical Neurological disease in children: A Global Epidemiological Assessment (PANGEA) Investigators. PICU-Based Rehabilitation and Outcomes Assessment: A Survey of Pediatric Critical Care Physicians. Pediatr Crit Care Med. 2019 Jun;20(6):e274-e282. doi: 10.1097/PCC.0000000000001940. PMID 30946294
- [Derived] Fink EL, Beers SR, Houtrow AJ, Richichi R, Burns C, Doughty L, Ortiz-Aguayo R, Madurski CA, Valenta C, Chrisman M, Golightly L, Kiger M, Patrick C, Treble-Barna A, Pollon D, Smith CM, Kochanek P; PICU-Rehabilitation Study Group. Early Protocolized Versus Usual Care Rehabilitation for Pediatric Neurocritical Care Patients: A Randomized Controlled Trial. Pediatr Crit Care Med. 2019 Jun;20(6):540-550. doi: 10.1097/PCC.0000000000001881. PMID 30707210